CLINICAL TRIAL: NCT02520726
Title: A Randomized, Double-blind, Placebo-controlled Pilot Study of Sertraline for the Prevention of PTSD in Burn Victims
Brief Title: PTSD Prevention Study Examining the Efficacy of Sertraline in Burn Victims
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Brent Kious, Psychiatry Resident, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UUtahIRB0062412
Record Dates: First submitted 2014-04-18; First posted 2015-08-13 (Estimated); Results first posted 2018-04-10 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2017-12

CONDITIONS: Post-traumatic Stress Disorder
Keywords: Posttraumatic stress disorder; PTSD; Sertraline; Burns
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Burns | interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sertraline (Experimental): Patients age 18-65: sertraline 50mg PO qday for one week, then 100mg PO qday for one week, then 150mg PO qday for one week, then 200mg PO qday for one week, with flexible titration. Patient age >65: sertraline 25mg PO qday for one week, then 50mg PO qday for one week, then 75mg PO qday for one week, then 100mg PO qday for one week, with flexible titration
  Interventions: Drug: Sertraline
- Placebo (Placebo Comparator): Placebo 1 capsule PO qday for one week, then 2 capsules PO qday for one week, then 3 capsules PO qday for one week, then 4 capsules PO qday for one week.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Sertraline — < 65years: sertraline 50mg PO qday increasing by 50mg per day per week until 200mg for one week, then stop.
  Other Names: Zoloft
  Arms: Sertraline
Drug: Placebo oral capsule — Matched encapsulated placebo from 1-4 capsules daily
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled study to determine whether administration of sertraline to patients who exhibit acute stress disorder secondary to severe burns can contribute to the prevention of post-traumatic stress disorder (PTSD).

ELIGIBILITY:
Inclusion Criteria:

* Victim of a traumatic event leading to personal injury
* Patient experienced a feeling of intense fear, hopelessness, or horror during the course of the event or immediately afterward
* Positive screen on the ASDS (for inclusion in the randomization phase); a total ASDS score of ≥ 37 (including a dissociative score of ≥ 9) will be counted as a positive screen.

Exclusion Criteria:

* Age < 18
* Pregnant women, lactating women, or women not using acceptable form of birth control
* Epilepsy or head trauma resulting in seizures
* Current or historical schizophrenia, bipolar disorder, mental retardation, OCD, eating disorders, dementia, delirium, or self-injurious behavior
* Current/previously diagnosed PTSD
* History of hypersensitivity to sertraline
* Trauma occurring > 7 days prior to likely first treatment in the randomization phase of the trial.
* Unable to provide informed consent for participation in the study protocol.
* Patient at high risk of recurrent bleeding despite surgical stabilization
* Patient with a history of serotonin syndrome
* Patient non-fluent in English
* Patient currently prescribed an antidepressant (any SSRI, SNRI, TCA, MAOI, mirtazapine, or trazodone in excess of 100mg per day)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brent M Kious, MD PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Hospital, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo 1 capsule PO qday for one week, then 2 capsules PO qday for one week, then 3 capsules PO qday for one week, then 4 capsules PO qday for one week.
  Sertraline: < 65years: sertraline 50mg PO qday increasing by 50mg per day per week until 200mg for one week, then stop.
Period: Overall Study
Arm/Group | Sertraline | Placebo
Started | 3 | 2
Completed | 0 | 0
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sertraline | Placebo | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Clinician-Administered PTSD Scale
Time Frame: Month
Population: All subjects lost to follow-up
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Beck Scale for Suicide Ideation
Time Frame: 1 month
Population: All subjects lost to follow-up
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Sertraline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes